CLINICAL TRIAL: NCT05598788
Title: Development of a Microsampling Approach for Personalized Monitoring of Kinase Inhibitor Targeted Therapies
Brief Title: Microsampling Approach for Monitoring of Kinase Inhibitor Targeted Therapies
Acronym: MISTIK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC22_8962_MISTIK
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2022-10

CONDITIONS: Blood Concentrations of Nine Anti-cancer Drugs : Axitinib, Olaparib, regorafénib, Cabozantinib, Niraparib, Talazoparib, Palbociclib, Abemaciclib, Tucatinib
Keywords: ORAL CHEMOTHERAPIES; AT HOME THERAPEUTIC DRUG MONITORING; MICROSAMPLING STRATEGY; CONCENTRATION EFFECT RELATIONSHIP; PERSONALIZED MEDICINE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurement of drug concentrations — Measurement of anti-cancer drug concentrations using volumetric absorptive micro-sampling (VAMS) and venous blood sample
  Other Names: Micro-sampling

SUMMARY:
The MISTIK project aims at clinically validating the technique of oral anticancer drugs determination by volumetric absorptive micro-sampling and at comparing the results to measurements performed on venous samples.

DETAILED DESCRIPTION:
The International recommendations for the validation of DBS-based methods will be applied (Capiau et al, TDM, 2019) by including 40 patients per molecule of interest. Nine drugs will be monitored : axitinib, olaparib, regorafénib, cabozantinib, niraparib, talazoparib, palbociclib, abemaciclib, tucatinib.

Two samples will be collected from each patient, one by venous sampling and the second at the same time (approximately) using a capillary blood sample derived from a finger prick.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with one of the 9 drugs concerned by the study : axitinib, olaparib, regorafénib, cabozantinib, niraparib, talazoparib, palbociclib, abemaciclib, tucatinib
* person who does not object to their participation in the research

Exclusion Criteria:

* Adults subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with one of the 9 drugs concerned by the study : axitinib, olaparib, regorafénib, cabozantinib, niraparib, talazoparib, palbociclib, abemaciclib, tucatinib
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of venous blood vs VAMS concentrations | 1 day
  Comparison of drug concentrations measured from the venous blood samples with concentrations measured from VAMS

CONTACTS AND LOCATIONS:
Overall Officials: VERDIER Marie-Clemence, Principal Investigator — Rennes University Hospital
Locations (3):
- France (3):
  - Centre Eugène Marquis Unicancer, Rennes
  - Rennes University Hospital, Rennes
  - Institut de cancérologie Strasbourg Europe, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided